CLINICAL TRIAL: NCT01688258
Title: A Prospective, Open Labeled, Multicenter, Diagnostic Study on the Detection of T. Pallidum, H. Ducreyi and HSV Type 1 and 2 From Genital, Anal and Oropharyngeal Ulcers With a New Multiplex Real-time Polymerase Chain Reaction
Brief Title: New Multiplex Real-time PCR for Genital Ulcer Disease
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: GUD-PCR
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Genital Ulcer Disease (GUD)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Diagnostic swab

SUMMARY:
(i) To compare a new diagnostic PCR with established diagnostic procedures for T. pallidum (serology, dark field microscopy), H. ducreyi (cultivation), HSV types 1 and 2 (cultivation, PCR).

(ii) To assess the frequency of infections with T. pallidum, H. ducreyi and HSV types 1 and 2 in patients with genital, anal and oropharyngeal ulcers by a new PCR.

ELIGIBILITY:
Inclusion criteria:

* Patient with genital, anal or oropharyngeal ulcers
* Age minimum of 18 years.
* Informed consent must be obtained from each patient/control patient in written form prior to any study procedure.

Exclusion criteria:

* Antibiotic therapy within 2 weeks before the visit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with genital, anal or oropharyngeal ulcers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Bosshard, PhD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Glatz M, Juricevic N, Altwegg M, Bruisten S, Komericki P, Lautenschlager S, Weber R, Bosshard PP. A multicenter prospective trial to asses a new real-time polymerase chain reaction for detection of Treponema pallidum, herpes simplex-1/2 and Haemophilus ducreyi in genital, anal and oropharyngeal ulcers. Clin Microbiol Infect. 2014 Dec;20(12):O1020-7. doi: 10.1111/1469-0691.12710. Epub 2014 Jul 25. PMID 24909546